CLINICAL TRIAL: NCT02089152
Title: A Single-blind Stepped Wedge Cluster Randomized Controlled Behaviour Change Trial to Determine Effectiveness of Prevention Programme of Melioidosis in Diabetics in Ubon Ratchathani, Northeast Thailand
Acronym: PREMEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: MICRO1307
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2019-09

CONDITIONS: Melioidosis
Keywords: Diabetes; Melioidosis; stepped wedge trial; behaviour change; Education program
MeSH Terms: conditions — Melioidosis; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cluster A (Other): General education for prevention of diabetic complications in year 1, Melioidosis prevention education in years 2, 3 and 4.
  Interventions: Other: An educational programme for prevention of melioidosis
- Cluster B (Other): General education for prevention of diabetic complications in year 1 and 2, Melioidosis prevention education in year 3 and 4.
  Interventions: Other: An educational programme for prevention of melioidosis
- Cluster C (Other): General education for prevention of diabetic complications in year 1, 2 and 3, Melioidosis prevention education in year 4.
  Interventions: Other: An educational programme for prevention of melioidosis

INTERVENTIONS:
Other: An educational programme for prevention of melioidosis — The intervention will be randomly implemented at 10, 10 and 10 diabetic clinics at the end of years 1, 2 and 3, respectively. The education will be conducted using small group education, in which 20 to 25 participants at a time will attend group sessions conducted by the study team.

SUMMARY:
Study hypothesis:

Prevention programme for melioidosis can reduce incidences of overall hospitalization due to infectious diseases and due to culture-confirmed melioidosis in diabetic population in northeast Thailand

This study is a prospective single-blind multicentre stepped wedge cluster randomized controlled behaviour change trial in 9,000 diabetics in Ubon Ratchathani, northeast Thailand.

DETAILED DESCRIPTION:
Melioidosis is an infectious disease caused by soil-dwelling Gram-negative bacilli Burkholderia pseudomallei. The disease is highly endemic in northeast Thailand. Diabetes mellitus is the major underlying risk factor for melioidosis, occurring in more than 50% of all culture-proven melioidosis patients. The annual incidence of melioidosis in diabetes in northeast Thailand is currently 244 per 100,000, and the overall case fatality rate is about 40%. The number of people dying from melioidosis is now comparable to deaths from tuberculosis, and exceeds those from malaria, diarrheal illnesses and measles combined. Melioidosis is potentially preventable since infection occurs as a direct result of exposure to B. pseudomallei in the environment. Nonetheless, most of Thai people have never heard of melioidosis, there is currently no vaccine for melioidosis, and formal prevention guideline are lacking worldwide.

The investigators recently developed new guidelines for the prevention of melioidosis in Thailand; including avoidance of direct contact with soil or environmental water and use of protective gear if contact is necessary, consumption of bottled or boiled water only, and avoidance of direct contact with heavy rain and dust clouds.

The investigators aim to conduct a clinical trial to determine effectiveness of the proposed prevention programme of melioidosis. The investigators also predict that the prevention programme of melioidosis will also prevent other common infectious diseases with have similar routes of infection, such as leptospirosis and acute diarrhea. The outcome of the RCT will be crucial evidence for the Ministry of Public Health (MoPH) Thailand for their consideration of policy changes for the prevention of melioidosis countrywide.

The funder: Wellcome Trust. Grant reference number: 101103/Z/13/Z

Result:

Pubmed link: https://pubmed.ncbi.nlm.nih.gov/34170931/

PLoS NTD link: https://journals.plos.org/plosntds/article?id=10.1371/journal.pntd.0009060

DOI: https://doi.org/10.1371/journal.pntd.0009060

MedRxiv: https://www.medrxiv.org/content/10.1101/2020.12.18.20248448v1

ELIGIBILITY:
Inclusion Criteria:

* Male or female (Include pregnant women) , aged from 18 to 65 years old
* Diagnosed of diabetes according to American Diabetes Association 2013 as following

  * Fasting plasma glucose (FPG) ≥ 126 mg/dl or
  * HbA1C ≥ 6.5% or
  * 2 hour plasma glucose (PG) ≥ 200 mg/dl during an OGTT or
  * Classic symptoms of hyperglycaemia with a random PG ≥ 200 mg/dl
* Oriented and conversed normally
* Willingness to participate in the study, and written, informed consent obtained from patient

Exclusion Criteria:

* Confused or unable to communicate
* Diagnosed of melioidosis and has not completed oral-eradicative treatment for melioidosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9075 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Overall hospital admissions due to infectious diseases | Up to 4 years
  Infectious diseases will be determined by International Classification of Disease 10 (ICD10) defined by attending physicians.
Culture-confirmed melioidosis | Up to 4 years
  Culture-confirmed melioidosis is defined as presentation with clinical features of melioidosis in association with cultures from any clinical specimen positive for Burkholderia pseudomallei.

SECONDARY OUTCOMES:
Overall mortality | Up to 4 years
  Overall mortality is defined as death from all causes.
Overall melioidosis | Up to 4 years
  Overall melioidosis is defined as a combination of culture confirmed melioidosis and clinical melioidosis. Clinical melioidosis is defined as presentation with clinical features of melioidosis in association with cultures from all clinical specimens negative for Burkholderia pseudomallei.

CONTACTS AND LOCATIONS:
Overall Officials: Assist Prof. Direk Limmathurotsakul, M.D., Principal Investigator — Mahidol-Oxford Tropical Medicine Research Unit (MORU), Faculty of Tropical Medicine, Mahidol university, Thailand
Locations (1):
- Sappasithiprasong Hospital, Ubon Ratchathani, Thailand

REFERENCES:
- [Background] Limmathurotsakul D, Wongratanacheewin S, Teerawattanasook N, Wongsuvan G, Chaisuksant S, Chetchotisakd P, Chaowagul W, Day NP, Peacock SJ. Increasing incidence of human melioidosis in Northeast Thailand. Am J Trop Med Hyg. 2010 Jun;82(6):1113-7. doi: 10.4269/ajtmh.2010.10-0038. PMID 20519609
- [Background] Limmathurotsakul D, Peacock SJ. Melioidosis: a clinical overview. Br Med Bull. 2011;99:125-39. doi: 10.1093/bmb/ldr007. Epub 2011 May 9. PMID 21558159
- [Background] Currie BJ, Dance DA, Cheng AC. The global distribution of Burkholderia pseudomallei and melioidosis: an update. Trans R Soc Trop Med Hyg. 2008 Dec;102 Suppl 1:S1-4. doi: 10.1016/S0035-9203(08)70002-6. PMID 19121666
- [Background] Limmathurotsakul D, Dance DA, Wuthiekanun V, Kaestli M, Mayo M, Warner J, Wagner DM, Tuanyok A, Wertheim H, Yoke Cheng T, Mukhopadhyay C, Puthucheary S, Day NP, Steinmetz I, Currie BJ, Peacock SJ. Systematic review and consensus guidelines for environmental sampling of Burkholderia pseudomallei. PLoS Negl Trop Dis. 2013;7(3):e2105. doi: 10.1371/journal.pntd.0002105. Epub 2013 Mar 21. PMID 23556010
- [Background] Suputtamongkol Y, Hall AJ, Dance DA, Chaowagul W, Rajchanuvong A, Smith MD, White NJ. The epidemiology of melioidosis in Ubon Ratchatani, northeast Thailand. Int J Epidemiol. 1994 Oct;23(5):1082-90. doi: 10.1093/ije/23.5.1082. PMID 7860160
- [Background] Faa AG, Holt PJ. Melioidosis in the Torres Strait islands of far North Queensland. Commun Dis Intell Q Rep. 2002;26(2):279-83. doi: 10.33321/cdi.2002.26.26. PMID 12206383
- [Background] Limmathurotsakul D, Kanoksil M, Wuthiekanun V, Kitphati R, deStavola B, Day NP, Peacock SJ. Activities of daily living associated with acquisition of melioidosis in northeast Thailand: a matched case-control study. PLoS Negl Trop Dis. 2013;7(2):e2072. doi: 10.1371/journal.pntd.0002072. Epub 2013 Feb 21. PMID 23437412
- [Background] Limmathurotsakul D, Wongsuvan G, Aanensen D, Ngamwilai S, Saiprom N, Rongkard P, Thaipadungpanit J, Kanoksil M, Chantratita N, Day NP, Peacock SJ. Melioidosis caused by Burkholderia pseudomallei in drinking water, Thailand, 2012. Emerg Infect Dis. 2014 Feb;20(2):265-8. doi: 10.3201/eid2002.121891. PMID 24447771
- [Background] Wongsuvan N, Malasit M, Hongsuwan M, et al. Defining beliefs and environmental contraints on prevention of melioidosis in northeast Thailand. 2013. (manuscript under preparation)
- [Background] Limmathurosakul D, Lubell Y, Day N, Peacock N. Modelling the cost-effectiveness of strategies to prevent melioidosis in northeast Thailand. 2013. (manuscript under preparation)
- [Background] Chaowagul W, White NJ, Dance DA, Wattanagoon Y, Naigowit P, Davis TM, Looareesuwan S, Pitakwatchara N. Melioidosis: a major cause of community-acquired septicemia in northeastern Thailand. J Infect Dis. 1989 May;159(5):890-9. doi: 10.1093/infdis/159.5.890. PMID 2708842
- [Background] Leelarasamee A, Bovornkitti S. Melioidosis: review and update. Rev Infect Dis. 1989 May-Jun;11(3):413-25. doi: 10.1093/clinids/11.3.413. PMID 2665001
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Cheng AC, Currie BJ, Dance DAB, Funnell SGP, Limmathurotsakul D, Simpson AJH, Peacock SJ. Clinical definitions of melioidosis. Am J Trop Med Hyg. 2013 Mar;88(3):411-413. doi: 10.4269/ajtmh.12-0555. PMID 23468355
- [Background] Moulton LH, Golub JE, Durovni B, Cavalcante SC, Pacheco AG, Saraceni V, King B, Chaisson RE. Statistical design of THRio: a phased implementation clinic-randomized study of a tuberculosis preventive therapy intervention. Clin Trials. 2007;4(2):190-9. doi: 10.1177/1740774507076937. PMID 17456522
- [Background] Hayes RJ, Bennett S. Simple sample size calculation for cluster-randomized trials. Int J Epidemiol. 1999 Apr;28(2):319-26. doi: 10.1093/ije/28.2.319. PMID 10342698
- [Background] Bursac Z, Gauss CH, Williams DK, Hosmer DW. Purposeful selection of variables in logistic regression. Source Code Biol Med. 2008 Dec 16;3:17. doi: 10.1186/1751-0473-3-17. PMID 19087314
- [Derived] Suntornsut P, Teparrukkul P, Wongsuvan G, Chaowagul W, Michie S, Day NPJ, Limmathurotsakul D. Effectiveness of a multifaceted prevention programme for melioidosis in diabetics (PREMEL): A stepped-wedge cluster-randomised controlled trial. PLoS Negl Trop Dis. 2021 Jun 25;15(6):e0009060. doi: 10.1371/journal.pntd.0009060. eCollection 2021 Jun. PMID 34170931